CLINICAL TRIAL: NCT01101373
Title: Bilateral Anterior Capsulotomy For Intractable Depression
Brief Title: Treatment of Severe Depressive Illness by Targeted Brain Surgery
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Trevor Hurwitz, Principal Investigator, University of British Columbia
Other Study IDs: H10-00851
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Major Depressive Disorder
Keywords: Limbic surgery; Stereotactic surgery; Major Depressive Disorder: Treatment Refractory
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All subjects who received BAC for treatment resistant depression between 2000 and 2009

SUMMARY:
This study will report on the outcome of a clinical program, operational since 1998, that has used surgery targeting an emotional pathway in the brain in the treatment of severe depressive illness that has failed to respond to all other available interventions. Benefit from surgery was anticipated on the basis that the lesion (bilateral anterior capsulotomy) is a well established surgical target for treating severe treatment resistant depression.

DETAILED DESCRIPTION:
Since 1998 bilateral anterior capsulotomy (BAC) has been available to patients in British Columbia Canada who have treatment refractory severe depressive illness. This study will report on the outcome of patients who have received this intervention. BAC is achieved by stereotactic radiofrequency lesioning. To date 8 patients have received BAC. For all patients there is follow-up data of at least 24 months. The purpose of this retrospective study is to report on the surgical protocol and to demonstrate the efficacy and safety of BAC in severe depression.

ELIGIBILITY:
Inclusion Criteria:

* Severe treatment resistant depression of at least 5 years duration
* older than 18 years

Exclusion Criteria:

* Comorbid organic mental disorder
* Delusional disorder
* Substance disorder
* Neurological disease
* Cluster B personality disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who received BAC for treatment resistant depression between 2000 and 2009
Sampling Method: Non-Probability Sample
Dates: Start 2000-10; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Honey, MD, Study Director — University of British Columbia; Judy Allen, MD, Study Director — University of British Columbia; Robert Hewko, MD, Study Director — University of British Columbia; Caroline Gosselin, MD, Study Director — University of British Columbia; Nicolas Bogod, MD, Study Director — University of British Columbia; Jeff Martzke, MD, Study Director — University of British Columbia; Patricia Taylor, Study Director — University of British Columbia
Locations (1):
- UBC Hospital, 2255 Wesbrook Mall, Vancouver, British Columbia, Canada